CLINICAL TRIAL: NCT06890819
Title: The Effect of Structured Feedback on Learning, Clinical Confidence and Anxiety in Psychiatric Nursing Students
Brief Title: The Effect of Structured Feedback on Learning, Clinical Confidence and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Tuba Çömez İkican, Tuba Çömez İkican, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024/434
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Structured Feedback; Clinical Decision-Making, Anxiety, Self-Confidence; Undergraduate Nursing Education; Learning Motivation
Keywords: Structured Feedback; Clinical Decision-Making, Anxiety, Self-Confidence; Undergraduate nursing education; Nursing Students; Learning motivation
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Experimental group (Experimental): Experimental: Experimental group
  Interventions: Behavioral: Assigned Interventions

INTERVENTIONS:
Behavioral: Assigned Interventions — Behavioral: Structured Feedback, Clinical Decision-Making, Anxiety, Self-Confidence,

SUMMARY:
This research is carried out by Dr Tuba Çömez İkican, and Dr. Olga İncesu. This research aimed to determine the effect of structured written and oral feedback given to students taking psychiatric nursing course on students' learning, self-confidence in clinical decision making and anxiety levels.

H1: Structured feedback significantly increases the learning level of nursing students. H2: Structured feedback increases nursing students' self-confidence in clinical decision--making. H3: Structured feedback decreases the level of anxiety felt by nursing students in the clinical decision-making process.The population of the study consisted of 3rd year students (N=52) studying in a Faculty of Nursing in the 2024-2025 academic year and performing the clinical practice of the Psychiatric Nursing course in a public hospital. After the purpose of the study was explained to the participants, all students (n=51) who met the criteria and gave written and verbal consent to participate in the study were included in the sample group. In the post hoc power analysis of the study, it was determined that the effect size (d)=0.85, α=0.05, the total sample size was 51, the power analysis result was 0.97 and the sample size was sufficient.

The research is a quasi-experimental research design with pre-test / post-test control.

Inclusion Criteria

* To be enrolled in the psychiatric nursing course,
* To be 18 years of age or older,
* To agree to participate in the research,
* To be able to perform the clinical practice of psychiatric nursing course,
* To continue clinical practice.

Data collected with the 'Personal Information Form', 'Self-Regulated Learning Scale for Clinical Nursing Practices', 'Self-confidence and Anxiety Scale for Clinical Decision Making in Nursing', 'Feedback Form' and 'Feedback Evaluation Form'

Institutional permission from Istanbul University School of Nursing and ethics committee approval (Number:04.12.2024-3050772) from Istanbul University Social and Human Sciences Research Ethics Committee obtained in order to conduct the study. Statistical analysis of research data will be done using a package program called SPSS (IBM SPSS Statistics 29). The expenses of the research will be covered by the researcher.

DETAILED DESCRIPTION:
Feedback, in the most general sense, refers to the reactions or responses received or given regarding an event, action or situation. The concept of feedback is very important in the field of education. When the studies on feedback in the national and international literature are examined, it has been determined that effective feedback contributes to students' evaluation of their performance, increasing self-regulated learning and seeing areas of development. Nursing education is a process that includes theoretical and practical teaching and learning, requires the acquisition of theoretical knowledge and manual skills, and requires observation and comment. During this process, students sometimes experience various difficulties, and this cause difficulties in learning and causes feelings of anxiety and lack of confidence in decision-making in the clinical field. A study in the field of nursing has shown that while written feedback allows students to see their deficiencies in their knowledge and skills, verbal feedback provides a faster response and offers the advantage of instant intervention in the learning process. However, there are various studies on how the quality of the feedback given during the feedback process of nursing students shapes students' confidence in clinical skills. Gillespie and Peterson (2009) state that verbal feedback allows students to ask questions more comfortably and encourages their active participation in the learning process. Written feedback, on the other hand, provides students with the opportunity to re-evaluate certain mistakes and think deeply about their learning process, thus contributing to students' long-term knowledge acquisition and improving their self-confidence and reducing their anxiety. In this context, this study was planned to determine the effects of verbal and written feedback given to students on students' learning, self-confidence in clinical decision-making, and anxiety levels.

This research aimed to determine the effect of structured written and oral feedback given to students taking psychiatric nursing course on students' learning, self-confidence in clinical decision making and anxiety levels.

H1: Structured feedback significantly increases the learning level of nursing students. H2: Structured feedback increases nursing students' self-confidence in clinical decision--making. H3: Structured feedback decreases the level of anxiety felt by nursing students in the clinical decision-making process.The population of the study consisted of 3rd year students (N=52) studying in a Faculty of Nursing in the 2024-2025 academic year and performing the clinical practice of the Psychiatric Nursing course in a public hospital. After the purpose of the study was explained to the participants, all students (n=51) who met the criteria and gave written and verbal consent to participate in the study were included in the sample group. In the post hoc power analysis of the study, it was determined that the effect size (d)=0.85, α=0.05, the total sample size was 51, the power analysis result was 0.97 and the sample size was sufficient.

The research is a quasi-experimental research design with pre-test / post-test control.

Dependent Variables: Self-Regulated Learning Scale for Clinical Nursing Practices score, Self-confidence and Anxiety Scale for Clinical Decision Making in Nursing score Independent Variables: Sociodemographic characteristics of the participants

Inclusion Criteria

* To be enrolled in the psychiatric nursing course,
* To be 18 years of age or older,
* To agree to participate in the research,
* To be able to perform the clinical practice of psychiatric nursing course,
* To continue clinical practice.

The study was conducted at Istanbul University Faculty of Nursing between December 2024- January 2025. Data will be collected through the "Personel Information Form", 'Self-Regulated Learning Scale for Clinical Nursing Practices', 'Self-confidence and Anxiety Scale for Clinical Decision Making in Nursing', 'Feedback Form' and 'Feedback Evaluation Form' The personal information form was prepared by the researchers in line with the literature. Permission was obtained from the scale owners for the scales to be used in the study.

* Socio-Demographic Characteristics Form: This form consists of a total of 7 questions including socio-demographic characteristics created by researchers within the framework of the literature.
* Self-Regulated Learning Scale for Clinical Nursing Practices: The scale was first developed by Satoko Iyama and Hitomi Maeda in 2017. Its Turkish validity and reliability were carried out by Şenol and Orgun in 2018. The scale is a 5-point Likert type. It consists of 16 items and 2 sub-dimensions, "Motivation" and "Learning Strategies". A minimum score of 16 and a maximum score of 80 can be obtained from the entire scale, and Cronbach α was found to be = 0.898.
* Self-Confidence Anxiety Scale for Clinical Decision Making in Nursing (HKKÖAÖ): The scale was first developed by White (2013). Its Turkish validity and reliability were carried out by Bektaş et al. (2015). The scale was developed to evaluate the anxiety and self-confidence levels of nursing students in clinical decision making and separate scores are obtained for self-confidence and anxiety. The scale consists of a total of 27 questions and 3 sub-dimensions (using sources and listening fully to obtain information, using available information to determine the problem, knowing and taking action). The increase in scores from self-confidence and its sub-dimensions indicates that students' self-confidence levels in clinical decision making have increased. Low scores from the anxiety section and its sub-dimensions indicate low anxiety levels in clinical decision making. It is a six-point (6) Likert-type scale. The lowest score that can be obtained from the self-confidence and anxiety sections is 27, and the highest score is 162. The total Cronbach's alpha of the self-confidence section of the scale was determined as 0.970; the total Cronbach's alpha of the anxiety section was determined as 0.969.
* Feedback Form: This form, which was created by the researchers in line with the literature, consists of a total of 3 questions regarding clinical practice and homework. - Feedback Evaluation Form: This form, created by researchers in line with the literature, consists of a total of 8 questions regarding the feedback given.

In the study, the data collection process began after obtaining ethics committee approval and institutional permission. Nursing students who meet the inclusion criteria will be identified, and data will be collected twice as pre-test and post-test. The data collection process is as follows:

Pre-intervention: Socio-Demographic Characteristics Form, Self-Regulated Learning Scale for Clinical Nursing Practices and Self-confidence and Anxiety Scale for Clinical Decision Making in Nursing will be administered as a pre-test to all students who give written and verbal consent to participate in the study and meet the inclusion criteria.

Intervention: The study will last for a total of 6 weeks. Firstly, written feedback will be given to the assignments given by the students every week with the Feedback Form prepared by the researchers. Afterwards (when the students' review of these forms is completed), a single educator will conduct structured interviews with the students every week, which are planned to be at least 20 minutes in the clinical practice of the mental health and psychiatric nursing course. Within the scope of this interview, the educator will give verbal feedback on the student's clinical practice process and the homework (interview recording form and nursing care plan) given by the student each week. In addition, if the student has any questions based on the written feedback, they will be answered. The feedback will be based on the strengths and aspects that need to be developed regarding the student's interview with the patient, diagnosis, nursing care planning, implementation and evaluation skills.

Post-intervention: At the end of the 6th week, students will be administered the Feedback Evaluation Form, the Self-Regulated Learning Scale for Clinical Nursing Practices and the Self-confidence and Anxiety Scale for Clinical Decision Making in Nursing as a post-test.

Institutional permission from Istanbul University School of Nursing and ethics committee approval (Number:04.12.2024-3050772) from Istanbul University Social and Human Sciences Research Ethics Committee obtained in order to conduct the study. Statistical analysis of research data will be done using a package program called SPSS (IBM SPSS Statistics 29). The expenses of the research will be covered by the researcher.

ELIGIBILITY:
Inclusion Criteria:

* To be enrolled in psychiatric nursing course,
* To be 18 years of age or older,
* To agree to participate in the research,
* To be able to perform the clinical practice of psychiatric nursing course,
* To continue clinical practice.

Exclusion Criteria:

* Be less than 18 years old,
* Not knowing how to read, write and speak Turkish,
* Having any cognitive, sensory and spiritual problems,
* Not willing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2024-12-24 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | Baseline
  Personal Information Form: This form was created by the researchers within the framework of the literature and consists of 7 questions about the participants' descriptive characteristics (age, gender, and GPA) and feedback experiences (status of receiving feedback before, effects of feedback, etc.).
Self-Regulated Learning Scale for Clinical Nursing Practices: | Baseline
  - Self-Regulated Learning Scale for Clinical Nursing Practices: The scale was first developed by Satoko Iyama and Hitomi Maeda in 2017. Its Turkish validity and reliability were carried out by Şenol and Orgun in 2018. The scale is a 5-point Likert type. It consists of 16 items and 2 sub-dimensions, "Motivation" and "Learning Strategies". A minimum score of 16 and a maximum score of 80 can be obtained from the entire scale, and Cronbach α was found to be = 0.898.
Nursing Anxiety and Self-Confidence with Clinical Decision Making Scale (NASC-CDM) | Baseline
  - Nursing Anxiety and Self-Confidence with Clinical Decision Making Scale (NASC-CDM): The scale was first developed by Satoko Iyama and Hitomi Maeda in 2017. Its Turkish validity and reliability were carried out by Şenol and Orgun in 2018. The scale is a 5-point Likert type. It consists of 16 items and 2 sub-dimensions, "Motivation" and "Learning Strategies". A minimum score of 16 and a maximum score of 80 can be obtained from the entire scale, and Cronbach α was found to be = 0.898.

SECONDARY OUTCOMES:
- Self-Regulated Learning Scale for Clinical Nursing Practices: | 5 weeks
  - Self-Regulated Learning Scale for Clinical Nursing Practices: The scale was first developed by Satoko Iyama and Hitomi Maeda in 2017. Its Turkish validity and reliability were carried out by Şenol and Orgun in 2018. The scale is a 5-point Likert type. It consists of 16 items and 2 sub-dimensions, "Motivation" and "Learning Strategies". A minimum score of 16 and a maximum score of 80 can be obtained from the entire scale, and Cronbach α was found to be = 0.898.
- Nursing Anxiety and Self-Confidence with Clinical Decision Making Scale (NASC-CDM): | 5 weeks
  - Nursing Anxiety and Self-Confidence with Clinical Decision Making Scale (NASC-CD): The scale was first developed by White (2013). Its Turkish validity and reliability were carried out by Bektaş et al. (2015). The scale was developed to evaluate the anxiety and self-confidence levels of nursing students in clinical decision making and separate scores are obtained for self-confidence and anxiety. The scale consists of a total of 27 questions and 3 sub-dimensions (using sources and listening fully to obtain information, using available information to determine the problem, knowing and taking action). The increase in scores from self-confidence and its sub-dimensions indicates that students' self-confidence levels in clinical decision making have increased. Low scores from the anxiety section and its sub-dimensions indicate low anxiety levels in clinical decision making.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No